CLINICAL TRIAL: NCT04801875
Title: Effectiveness of the Selected Exercise Program on Non-specific Cervical Pain in Ney and Violin Performers
Brief Title: Cervical Pain and Exercise in Musicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/14
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cervical Pain
Keywords: Exercise; Cervical Pain; Disabilities; Musicians
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study was based on pre-test and post-test methods. Musicians who met inclusion criterion were assigned to violin and ney groups according to performing musical instrument.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Violin Performers (Experimental): Violin performers received three 40-45 minute exercise sessions each week for eight weeks. The selected exercise program designed to correct postural alignment.
  Interventions: Other: Selected Exercise
- Ney Performers (Experimental): Ney performers received three 40-45 minute exercise sessions each week for eight weeks. The selected exercise program designed to correct postural alignment.
  Interventions: Other: Selected Exercise

INTERVENTIONS:
Other: Selected Exercise — The violin and ney groups performed a structured exercise training program 3 times a week for a total of 8 weeks. Adherence to the exercise training program was checked using a follow-up schedule to ensure regular participation of the musicians. The 8-week exercise training program was given with same physiotherapist under the same conditions. The every exercise session consisted of warm-up (3-5 min), main exercise (30-35 min) and cooling periods (3-5 min). The main exercise period was included ROM (10 min), stretching (5-7 min), isometric (5-10 min) and stabilization exercises (5 min).

SUMMARY:
Exercise training that is one of the effective treatment methods for cervical pain, is crucial in developing mobility and stability. Exercise training significantly reduces cervical pain as it advances postural alignment and neuromuscular coordination. In many single group studies on cervical pain in violin performers, it has been reported that the stabilization exercises have favorable consequences on pain relief and postural correction. But, there are no studies comparing ney and violin performers and analyzing the effectiveness of exercise training on non-specific cervical pain. The aim of this study is to search the effects of selected exercise training on pain, disability, range of motion, flexibility, strength and quality of life in ney and violin performers with non-specific cervical pain.

ELIGIBILITY:
Inclusion Criteria:

* Being professional musicians
* Using violin or ney musical instruments
* Had non-specific cervical pain during 3 months

Exclusion Criteria:

* Had cervical surgery in the last 3 months, discogenic pain, radiculopathy, neurological or systemic disorders,
* Missing exercise training session more than 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  Visual Analog Scale (VAS) was used to measure the severity of pain. In this scale, "0" indicates no pain, "10" indicates the highest value for perceived pain. Participants were asked to illustrate the intensity of the pain they felt on a material with a horizontal line of 10 cm and was recorded as VAS score.
Functional Status | 8 weeks
  The Northwick Park Neck Pain Questionnaire (NPQ) was used to specify functional status. NPQ was developed to designate the level of disability in neck pain; It is a 9-item scale including neck pain severity, neck pain and sleep, numbness and tingling in the arms at night, duration of symptoms and complaints, weight-bearing, reading and watching television, work and housework, social activities, and driving. It evaluates the severity, symptoms, duration of neck pain and disability in the activities specified in each item. Each of them consists of 5 items and is scored between 0-4 points. Neck pain total score consists of 36 points. If the patients are not driving, the total score is calculated over 32 points.
Life Quality | 8 weeks
  Quality of life was evaluated with the SF-36 scale. The scale consists of 8 sub-parameters with a total of 36 items. These sub-parameters are listed as; physical function, physical role limitation, pain, general health, energy (vitality), social function, emotional role limitation and mental health.

SECONDARY OUTCOMES:
Muscle Strength | 8 weeks
  Muscle strength was measured with a digital muscle dynamometer (Jtech Commander Muscle Testing). Anterior and middle part of deltoid, serratus anterior, upper and middle part of trapezius, cervical flexor and extensor muscles were measured.
Grip Strength | 8 weeks
  The grip strength was measured with a hand dynamometer (Baseline, Hydraulic Hand Dynamometer). Measurements were made in a sitting position, regardless of the right or left hand, with the elbow flexed at 90° and the arms in contact with the body without any abduction movement. In this position, Individuals were asked to squeeze their hand with maximum force and measurements were repeated for other arm.
Range of Motion | 8 weeks
  Cervical Flexion, extension, rotation and lateral flexion were measured by using a universal goniometer. Head and trunk were held upright while participants were in a sitting position.
Spinal Mobility | 8 weeks
  The jaw-sternum and jaw-wall distance were measured with a tape measure. Participants was asked to stand upright in an anatomical position while leaning against the wall. In this position, the distance of chin tip to wall and chin tip to the incisura jugularis were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan kalyoncu üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan C, Driscoll T, Ackermann B. Development of a specific exercise programme for professional orchestral musicians. Inj Prev. 2013 Aug;19(4):257-63. doi: 10.1136/injuryprev-2012-040608. Epub 2012 Dec 4. PMID 23211353
- [Background] Kuo YL, Lee TH, Tsai YJ. Evaluation of a Cervical Stabilization Exercise Program for Pain, Disability, and Physical Impairments in University Violinists with Nonspecific Neck Pain. Int J Environ Res Public Health. 2020 Jul 28;17(15):5430. doi: 10.3390/ijerph17155430. PMID 32731521
- [Background] Ackermann B, Driscoll T, Kenny DT. Musculoskeletal pain and injury in professional orchestral musicians in Australia. Med Probl Perform Art. 2012 Dec;27(4):181-7. PMID 23247873